CLINICAL TRIAL: NCT04822168
Title: Effects of Remote Motivational Enhancement & MySafeRx on Post-Detox Engagement and Retention in B/N Treatment (MySafeRx) - RCT
Brief Title: Effects of Remote Motivational Enhancement & MySafeRx on Post-Detox Engagement in B/N Treatment -RCT
Acronym: MySafeRx
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not implemented due to. change in study site and scope.
Sponsor: University of South Florida (Other)
Collaborators: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038163 - RCT
Record Dates: First submitted 2020-02-27; First posted 2021-03-30 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Care (Active Comparator): Standard Care through detox-based opioid treatment with B/N and weekly urine toxicology screening
  Interventions: Other: Standard Care
- MySafeRx™ Intervention (Experimental): The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of B/N medication within a secure medication storage device, and a standardized protocol for supervising self-administration of medication via videoconferencing.
  Interventions: Other: MySafeRx™

INTERVENTIONS:
Other: MySafeRx™ — The MySafeRx™ platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of B/N medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing.
  Arms: MySafeRx™ Intervention
Other: Standard Care — Standard Care through office-based opioid treatment with B/N dosing, on-site counseling and regular urine toxicology screening
  Arms: Standard Care

SUMMARY:
Opioid overdoses are a significant problem nationwide and novel interventions that can prevent overdose by improving Buprenorphine/ Naloxone (B/N) treatment for opioid use disorder are a public health priority. This study will both investigate the effects of starting remote motivational enhancement during inpatient detoxification on rates of engagement in B/N treatment and evaluate the impact of MySafeRx, a mobile device application which integrates remote motivational coaching with daily observed dosing from secure electronic pill dispensers at home via videoconference, on treatment retention and overdose prevention. Broad dissemination of this new intervention could help communities across the nation expand and advance their capacity to increase B/N treatment engagement and retention, enhance medication adherence, and prevent overdose.

DETAILED DESCRIPTION:
The objective of this study is to conduct a randomized controlled trial (RCT) to evaluate an innovative strategy among opioid use disorder patients being discharged from detox. This study will evaluate the extent to which remote motivational enhancement sessions via videoconference and the option for flexible daily dosing at home with MySafeRx can improve engagement and retention with B/N treatment after detox in a county where access to outpatient, take-home B/N prescriptions are more limited compared to in-person daily B/N dosing and treatment. This study seeks to expand our understanding about what works to prevent opioid overdose by incorporating a RCT evaluating the effects of remote motivational enhancement (RME) sessions provided via videoconferencing at an inpatient detox facility and during early treatment in order to increase treatment engagement with daily outpatient supervised-dosing of B/N. Participants will use an Android smartphone device to access the MySafeRx app and complete their daily motivational interview sessions. This study will generate new knowledge about the most effective way to prevent overdose and engage patients in B/N treatment with observed daily dosing.

The primary aim of this study is:

Engagement: To examine the effect of Remote Motivational Enhancement (RME) sessions + MySafeRx Inspire Flex versus information alone + ACTS Standard Care on early engagement in outpatient B/N treatment based on the number of daily doses of prescribed B/N during the first 5 weeks post-detox.

Hypothesis: Participants enrolled in RME + MySafeRx Inspire Flex arm will be engaged in outpatient B/N treatment with significantly higher number of daily doses of prescribed B/N during the first 5 weeks post-detox than the information alone arm.

Secondary Aims:

Early Engagement: To examine the effect of RME + MySafeRx Inspire Flex versus information alone + ACTS Standard Care B/N treatment on early engagement in B/N treatment based on the proportion of participants a) who receive at least one outpatient B/N dose in first 7 days and b) who receive at least one outpatient B/N prescription at ACTS in the first 14 days post discharge from detox.

Opioid-Related Deaths: To examine the effects of RME + MySafeRx Inspire Flex versus information + ACTS Standard Care B/N on number of opioid-related deaths (as measured by county coroner report and clinic report) during the 6-months after discharge from inpatient detox.

Opioid Use (toxicology): To examine the differences in opioid use as measured by monthly urine toxicology for illicit opioids between MySafeRx Inspire Flex and information alone + ACTS Standard Care B/N treatment during a 24-week study period.

Other Pre-Specified Outcomes:

Overdoses: To examine the effect of RME + MySafeRx Inspire Flex versus information + ACTS Standard Care B/N treatment on the number of self-reported (with and without naloxone administered), county coroner reported, and clinic-reported opioid overdoses, throughout the 24 weeks of the study follow-up.

Opioid Use (self-report): To examine the differences in self-reported illicit opioid use between MySafeRx Inspire Flex information alone + ACTS Standard Care B/N treatment.

Treatment Retention: To examine the effect of RME + MySafeRx Inspire Flex versus information alone + ACTS Standard Care on retention in B/N treatment based on active B/N prescription at 12 and 24-week period.

Mental Health Symptoms: To examine the differences in mental health symptomatology using the BSI between MySafeRx Inspire Flex versus information alone + ACTS Standard Care B/N treatment during the 24-week study period.

For the current proposal, the investigators plan to recruit up to 120 B/N eligible patients during the high-risk period of transition out of detox into outpatient B/N treatment in order to be able to randomize 104 participants. Study participants will be recruited from the outpatient detox program at ACTS in Tampa, Florida. The investigators aim to recruit 2 patients a week for the study and randomize, on average, one patient to the MySafeRx program each week. Study participants will participate in a baseline assessment and six follow-up assessments at week 4, week 8, week 12, week 16, week 20, and week 24. These assessments will be conducted by the project coordinator and will occur via phone or at the ACTS facility (baseline assessment will always occur at ACTS detox prior to discharge). To protect the privacy of this information, the assessments will be identified only by a code number linked to study participants with a key that is only accessible to the data analyst. Study assessments will take approximately one and a half hours to complete.

Once the participant has consented, completed the baseline assessment, and a PI or Co-I has approved them to participate, they will be randomized to either MySafeRx or Standard Care. Given the study population, the investigators assume there will be some loss of participants at follow-up. The investigators have planned for this in the assessment of appropriate sample size, as well as in the data analysis procedures.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* opioid use disorder
* stepping down from inpatient detox services
* willing to engage in daily outpatient supervised dosing of B/N.

Exclusion Criteria:

* cognitively impaired (Unable to complete consent quiz at 90% accuracy AND MOCA < 25/30 relative exclusion requiring PI approval, absolute exclusion for MOCA<21/30) (Nasreddine,et al., 2005)
* homeless without any expressed interest in attaining housing after detox discharge
* reporting active homicidal or suicidal ideation with an imminent plan
* current mania or psychosis
* expected incarceration in next 3 months (those that are incarcerated during the study will be removed from the study)
* unable or unwilling to use a mobile device
* medical contraindication to B/N
* unable to complete baseline assessments
* unstable medical illness who expect hospitalization in the next 3 months
* pregnant women (if a patient becomes pregnant while participating in this study, they will be withdrawn)
* prisoners
* court-ordered individuals
* is non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-04-05 (Estimated); Study Completion 2022-04-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Remote Motivational Enhancement (RME) Sessions on Early Engagement in B/N Treatment | 5 weeks
  To examine the effect of Remote Motivational Enhancement (RME) sessions + MySafeRx Inspire Flex versus information alone + ACTS Standard Care on early engagement in outpatient B/N treatment based on the number of daily doses of prescribed B/N during the first 5 weeks post-detox.

SECONDARY OUTCOMES:
Proportion of days engaged in dosing of B/N during first 2 weeks. | 2 weeks post discharge
  To examine the effect of RME + MySafeRx Inspire Flex versus information alone + ACTS Standard Care B/N treatment on early engagement in B/N treatment based on the proportion of participants a) who receive at least one outpatient B/N dose in first 7 days and b) who receive at least one outpatient B/N prescription at ACTS in the first 14 days post discharge from detox.
Opioid-Related Deaths | 24 weeks
  To examine the effects of RME + MySafeRx Inspire Flex versus information + ACTS Standard Care B/N on number of opioid-related deaths (as measured by county coroner report and clinic report) during the 6-months after discharge from inpatient detox.
Illicit Opioid Use Measured by Urine Toxicology Screening | 24 weeks
  To examine the differences in opioid use as measured by monthly urine toxicology for illicit opioids between MySafeRx Inspire Flex and information alone + ACTS Standard Care B/N treatment during a 24-week study period.

OTHER OUTCOMES:
Number of Opioid Overdoses (Total of non-fatal self-report, clinic-reported, and fatal) | 24 weeks
  To examine the effect of RME + MySafeRx Inspire Flex versus information + ACTS Standard Care B/N treatment on the number of self-reported (with and without naloxone administered), county coroner reported, and clinic-reported opioid overdoses, throughout the 24 weeks of the study follow-up.
Self-Reported Opioid Use | 24 Weeks
  To examine the differences in self-reported illicit opioid use between MySafeRx Inspire Flex information alone + ACTS Standard Care B/N treatment.
Outpatient Buprenorphine Treatment Retention | 24 Weeks
  To examine the effect of RME + MySafeRx Inspire Flex versus information alone + ACTS Standard Care on retention in B/N treatment based on active B/N prescription at 12 and 24-week period.
Mental Health Symptomatology | 24 weeks
  To examine the differences in mental health symptomatology using the BSI between MySafeRx Inspire Flex versus information alone + ACTS Standard Care B/N treatment during the 24-week study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, PhD, Principal Investigator — University of South Florida; Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- ACTS Adult Addiction Receiving Facility (AARF), Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to our outcome measures will be included in the IPD sharing plan, in addition to our study protocol, informed consent, and analytic plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and within 12 months of completion of the analysis of study primary aims, anonymous and de-identified data will be made available at the Open Science Framework (http://osf.io/) and/or Harvard Dataverse (https://dataverse.harvard.edu/) so that other investigators can verify or follow-up on the reported analyses.
Access Criteria: Anonymous and de-identified data will be stored on the Open Science Framework website (http://osf.io/) and/or Harvard Dataverse to be made available to other researchers to verify the research results. Before publication, only USF and CHA investigators will have direct access to the data, and only the CHA HERLab investigators will have access to the analyses.

REFERENCES:
- [Background] Schuman-Olivier Z, Borodovsky JT, Steinkamp J, Munir Q, Butler K, Greene MA, Goldblatt J, Xie HY, Marsch LA. MySafeRx: a mobile technology platform integrating motivational coaching, adherence monitoring, and electronic pill dispensing for enhancing buprenorphine/naloxone adherence during opioid use disorder treatment: a pilot study. Addict Sci Clin Pract. 2018 Sep 24;13(1):21. doi: 10.1186/s13722-018-0122-4. PMID 30249279

DOCUMENTS (1):
  • Informed Consent Form (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT04822168/ICF_000.pdf